CLINICAL TRIAL: NCT00372372
Title: The Efficacy of Risedronate in Prevention of Bone Loss in Patients Receiving High Dose Corticosteroid Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HARECCTR0500019
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2007-09-28 (Estimated); Status verified 2007-09

CONDITIONS: Osteoporosis
Keywords: corticosteroids, bone mineral, risedronate, bisphosphonate
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: risedronate

SUMMARY:
The efficacy of risedronate in prevention of bone loss in patients receiving high dose corticosteroid treatment

DETAILED DESCRIPTION:
We compare the effect of risedronate with placebo in bone mineral density changes in patients receiving high dose corticosteroids for their underlying diseases

ELIGIBILITY:
Inclusion Criteria:

1. Patients with various medical conditions who require high dose glucocorticoid treatment: (1) pulse methylprednisolone; (2) oral prednisolone (>=0.8mg/kg/day) or equivalent for at least 6 weeks.
2. Age>=18 years and <75 years.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Uncorrected hypocalcemia.
3. History of esophageal stricture.
4. Previous intolerance or hypersenstivity to biphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
bone mineral density

SECONDARY OUTCOMES:
Adverse events, new vertebral fractures

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD FRCP, Principal Investigator — Tuen Mun Hospital Hong Kong
Locations (1):
- Tuen Mun Hospital, Hong Kong, China